CLINICAL TRIAL: NCT06015347
Title: The Relationship Between Motor Development Between 1-18 Months and the Risk of Developmental Coordination Disorder (DCD) in the Preschool Period and Cerebral Palsy (CP) in Risky Infants
Brief Title: The Relationship Between Developmental Level in Infancy and Preschool Motor Performance in Risky Infants
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ozge Karanlik, Msc, Marmara University
Other Study IDs: MU-FTR-OK-01
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy; Developmental Coordination Disorder
Keywords: Cerebral Palsy; Developmental Coordination Disorder; Infant, Premature; Child Development
MeSH Terms: conditions — Cerebral Palsy; Motor Skills Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment: Infants at risk rated with the Alberta Infant Motor Scale between 1-18 months

SUMMARY:
The primary purpose of this study is to evaluate the relationship between the developmental level between 1-18 months and gross motor performance in the preschool period in risky infants followed up from a center for early intervention, and to determine the risk of developmental coordination disorder in the preschool period in risky infants.Gross Motor Function Measurement-88 will be applied to children diagnosed with cerebral palsy in the pre-school period to evaluate motor performance, among risky infants evaluated by Alberta Infant Motor Scale between 1-18 months.

Developmental Coordination Disorder Questionnaire will be applied to healthy children in order to evaluate the risk of gross motor performance and developmental coordination disorder.

DETAILED DESCRIPTION:
Risky infants are at risk in terms of development. Cerebral palsy, mental retardation, visual and hearing disorders are seen as major neurodevelopmental disorders, developmental coordination disorder, attention deficit and hyperactivity disorder and learning disability are seen as minor. In order to detect major and minor disorders that may be seen in the future, these infants should be evaluated periodically in terms of neurodevelopment from birth.There are many reliable tests in the neurodevelopmental evaluation of risky infants, and one of them is the Alberta Infant Motor Scale.

Alberta Infant Motor Scale (AIMS) assesses motor performance and level of development from birth to 18 months. AIMS finds a total of 58 items in 4 different positions, and each item is 1 point. The scores obtained in all positions are added together and this score is converted into a percentile score that shows the baby's status relative to his/her peers. When looking at the norm chart of AIMS, there are 5%, 10%, 25%, 50%, 75%, and 90% lines. The 5% and 10% norm lines are used as cutoff lines for abnormal motor development.

Gross Motor Function Measure-88 is used to evaluate gross motor performance and function change in children aged 15 months to 13 years with cerebral palsy and Down syndrome. There are a total of 88 items in 5 categories (supine and prone 17, sitting 20, crawling and kneeling 14, standing 13, walking, running, and climbing stairs 24). Scoring is done according to the ability to perform gross motor functions correctly. Scoring is done in the range of 0 - 3. If he/she starts the activity, 0 points, 1 point if he/she starts the activity, 2 points if he/she completes the activity partially, and 3 points if he/she completes the activity independently. Categories and total scores are calculated as a percentage (%).

Developmental Coordination Disorder Questionnaire is a 15-item questionnaire used to measure developmental coordination disorder risk and evaluate motor performance and skills in children aged 5-15 years. It consists of 15 items. Scoring is between 1 and 5 (1 = not similar, 5 = very similar). The maximum score that can be obtained from the test is 75. The range of scores indicating the risk of developmental coordination disorder varies according to age. 5-7 years - 15-46 points; 8-9 years - 15-55 points; It means that there is a risk of DCD developmental coordination disorder between the ages of 10-15 - 15-57 points.

ELIGIBILITY:
Inclusion Criteria:

* To take part in the risky baby classification,
* Being between the ages of 4-6,
* To have been evaluated with the Alberta Infant Motor Scale at the Turkish Spastic Children Foundation Family Counseling Center,
* To agree to participate in the study and to have the informed consent form approved by the family.

Exclusion Criteria:

* The family does not approve the informed consent form,
* Not being evaluated with the Alberta Infant Motor Scale,
* Diagnosis of Down syndrome and genetic syndrome,
* Being outside the age range,
* Currently having a health problem that would prevent assessment.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: At-risk infants currently aged 4-6 years and evaluated with the Alberta Infant Motor Scale
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Developmental Coordination Disorder Questionnaire | 4-6 years
  Developmental Coordination Disorder Questionnaire is a 15-item questionnaire used to measure developmental coordination disorder risk and evaluate motor performance and skills in children aged 5-15 years. It consists of 15 items. Scoring is between 1 and 5 (1 = not similar, 5 = very similar). The maximum score that can be obtained from the test is 75. The range of scores indicating the risk of developmental coordination disorder varies according to age. 5-7 years - 15-46 points; 8-9 years - 15-55 points; It means that there is a risk of developmental coordination disorder between the ages of 10-15 - 15-57 points.

SECONDARY OUTCOMES:
Gross Motor Function Measure-88 | 4-6 years
  Gross Motor Function Measure-88 is used to evaluate gross motor performance and function change in children aged 15 months to 13 years with cerebral palsy and Down syndrome. There are a total of 88 items in 5 categories (supine and prone 17, sitting 20, crawling and kneeling 14, standing 13, walking, running, and climbing stairs 24). Scoring is done according to the ability to perform gross motor functions correctly. Scoring is done in the range of 0 - 3. If he/she starts the activity, 0 points, 1 point if he/she starts the activity, 2 points if he/she completes the activity partially, and 3 points if he/she completes the activity independently. Categories and total scores are calculated as a percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Ozge KARANLIK, Principal Investigator — Marmara University
Locations (1):
- Turkish Spastic Children Foundation, Istanbul, Atasehir, Turkey (Türkiye)